CLINICAL TRIAL: NCT01715376
Title: Prospective Cohort Study on Integrated Treatment by Traditional Chinese and Western Medicine of Patients Diagnosed as CHD (Coronary Heart Disease) With Stable Angina
Brief Title: Effects of Integrated Treatment by Traditional Chinese and Western Medicine in Reducing Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: Changchun University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, yue deng, Director of cardiology department, Changchun University of Chinese Medicine
Other Study IDs: 201007001-3-1
Record Dates: First submitted 2012-09-14; First posted 2012-10-29 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Angina Pectoris; Coronary Artery Disease; Coronary Disease; Heart Disease; Cardiovascular Disease; Chest Pain; Pain; Signs and Symptoms; Arteriosclerosis
Keywords: traditional chinese medicine; complementary therapies; traditional chinese medicine syndrome scale
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Chest Pain; Pain; Signs and Symptoms; Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Integrative Chinese and western medicine: Integrative Chinese and western medicine group treat with western medical therapy for CHD refering to the 'Chronic stable angina pectoris diagnosis and treatment guide'which is published by Chinese society of Cardiology, Chinese Medical Association in March, 2007, including the anti-ischemia treatment(nitric acid ester,β-blocker,calcium antagonist,ACEI), anti platelet therapy(aspirin and/or clopidogrel) and other statins.TCM should be confirmed by the physicians, according to the syndrome differentiation and the treat plan recommended in this study.
- Western medicine: western medical therapy for CHD can refer to the 'Chronic stable angina pectoris diagnosis and treatment guide'which is published by Chinese society of Cardiology, Chinese Medical Association in March, 2007, including the anti-ischemia treatment(nitric acid ester,β-blocker,calcium antagonist,ACEI), anti platelet therapy(aspirin and/or clopidogrel) and other statins.

SUMMARY:
Compared with standardized western medical drug therapy, this study is mainly about whether the combination of standardized western medical drug therapy and Chinese medical continued treatment, can further decrease the rate of cardiovascular events for stable angina patients and change the condition of angina.

DETAILED DESCRIPTION:
We will pick 1100 patients who are according with the II、III stage in CHD western medical diagnosis standard, treat them with combination of standardized western medical drug therapy and Chinese medical continued treatment, or only with standardized western medical drug therapy,the treat course will last 6 months. The patients will be separated in two groups: Integrative treatment of Chinese medicine and western medicine group(integrative group) and western medical group according to the exposure factors(whether the patients accept differentiation of TCM ) during the follow-up period, observe the main indexes: Primary Endpoint: all because of death, stroke, nonfatal myocardial infarction, revascularization. Secondary endpoint: the events needed hospitalization which are because of (acute coronary syndrome)ACS,heart failure, severe arrhythmia, and complications. Secondary indexes: angina symptoms. Including the attack times, lasting time, inducing factors of angina attacks, pain degree of angina, discontinue rate of nitroglycerin, and electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. the patients who are according with the II、III stage in CHD western medical diagnosis standard；
2. age between 18 and 75(including 18 and 75)；
3. Signed the informed consent voluntarily.

Exclusion Criteria:

1. The patients whose systolic pressure≥180mmHg and/or diastolic pressure≥110mmHg, have sever insufficiency of heart and lung（cardiac function﹥Ⅱdegree）, sever arrhythmia（rapid atrial fibrillation, atrial flutter,paroxysmal ventricular tachycardia and so on）；
2. the patients who have myocardial infarction or vascular remodeling in last 3 months；
3. hepatic and kidney function obstacle（ALT、AST>1.5 times of normal upper limit value）；
4. the patients who cannot control blood glucose properly（fasting blood glucose>7.0mmol/L and/ or random blood glucose>11.0mmol/L）；
5. the patients who have stroke in late 6 months（lacunar cerebral infarction is not included）；
6. any other sever diseases such as malignant tumor；
7. the patients who attending other clinical study in late 3 months；
8. pregnant or lactating women；
9. the patients who have allergic constitution or are allergic to many drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: treat with combination of standardized western medical drug therapy and Chinese medical continued treatment
Sampling Method: Probability Sample
Enrollment: 1042 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Primary end point all cause death | up to 12 months
  all because of death, stroke, nonfatal myocardial infarction, revascularization.
Secondary endpoint hospitalization | up to 12months
  the events needed hospitalization which are because of (acute coronary syndrome)ACS,heart failure, severe arrhythmia, and complications

SECONDARY OUTCOMES:
Angina symptoms | up to 12months
  Including the attack times, lasting time, inducing factors of angina attacks, pain degree of angina, discontinue rate of nitroglycerin.
electrocardiogram | up to 12months

OTHER OUTCOMES:
safety indicators | up to 12months
  ALT ,AST,BUN,CR,blood routine examination,urine routine

CONTACTS AND LOCATIONS:
Overall Officials: deng yue, Study Chair — dirctor
Locations (1):
- Jilin Province TCM Institute of Chinese Medicine, Changchun, Jilin, China